CLINICAL TRIAL: NCT04669015
Title: NOVATION-1: A Randomized, Double-Blind, Placebo-Controlled, Phase III Study to Evaluate the Safety and Efficacy of Aerosolized Novaferon + SOC vs. Placebo + SOC in Hospitalized Adult Patients With Moderate to Severe COVID-19
Brief Title: Phase 3 Inhaled Novaferon Study in Hospitalized Patients With Moderate to Severe COVID-19
Acronym: NOVATION-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genova Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JH-COR-003
Record Dates: First submitted 2020-12-14; First posted 2020-12-16 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Covid19
Keywords: antiviral; SARS-CoV-2; COVID19
MeSH Terms: conditions — COVID-19 | interventions — recombinant interferon alpha 2b-like protein; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active plus SOC (Experimental): Inhaled Novaferon, given 20 ug BID, daily for 10 days, plus Standard of Care
  Interventions: Biological: Novaferon
- Placebo plus SOC (Placebo Comparator): Inhaled vehicle formulation (placebo), given BID, daily for 10 days, plus Standard of Care
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Novaferon — a novel recombinant antiviral protein drug
  Other Names: Standard of Care
  Arms: Active plus SOC
Biological: Placebo — Formulation vehicle
  Other Names: Standard of Care
  Arms: Placebo plus SOC

SUMMARY:
This study is a randomized, double-blind, multicenter, placebo-controlled trial to evaluate the safety and efficacy of a novel therapeutic agent, Novaferon, in hospitalized adult patients diagnosed with COVID-19. The study is comprised of two cohorts:

* Cohort A: This is a blinded safety lead-in comprising two arms. 40 patients will be randomized on a 1:1 basis to receive either Novaferon or matched placebo via a commercial nebulizer, plus Standard of Care (SOC)
* Cohort B: This is the main portion of the study, which comprises two arms. Up to 874 patients will be randomized on a 1:1 basis to receive either Novaferon or matched placebo via a commercial nebulizer, plus SOC

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Signed informed consent form by any patient capable of giving consent, or, when the patient is not capable of giving consent, by his or her legal/authorized representatives prior to initiation of any study procedures.
2. Men and women, ≥18 years of age at time of enrollment.
3. Laboratory-confirmed diagnosis of SARS-CoV-2 infection as determined by PCR, or other health authority-approved commercial assay or other validated public health assay in any specimen within 72 hours prior to randomization (point-of-care viral infection test allowable if RT-PCR test result not available only at the time of screening).
4. Less than or equal to 9 days from COVID-19 symptom onset to starting treatment.

   • Symptoms are defined as one or more of the following: cough, fever, shortness of breath, chest pain, abdominal pain, nausea/vomiting, diarrhea, body aches, weakness/fatigue, chills/sweating, headache, confusion, sore throat, runny nose/congestion, loss of taste or smell, or any other COVID-19 symptoms as determined by the Investigator.
5. Hospitalized and i) requiring supplemental oxygen by face mask or nasal prongs, or ii) non-invasive ventilation or iii) high-flow oxygen (WHO category 4 or 5)
6. Female patients participating in this study must agree to avoid becoming pregnant and have a negative pregnancy test prior to randomization. Male and female patients of reproductive potential must use a highly effective, protocol-specified method of contraception during the study and up to post 30 days after the last dose of study drug. For a list of protocol-specified contraceptive methods, and the definition of reproductive potential, refer to Appendix 1.

Exclusion Criteria:

Exclusion Criteria:

1. Known hypersensitivity or intolerance to Interferon (IFN) or Novaferon or any excipient(s) of Novaferon, including pre-existing allergy or hypersensitivity to ampicillin.
2. Currently undergoing invasive mechanical ventilation (including venous ECMO).
3. Inability to use a nebulizer with a mouthpiece.
4. ALT/AST > 5 times the Upper Limit of Normal (ULN) or a history of decompensated cirrhosis.
5. Stage 4 severe chronic kidney disease or requiring dialysis (i.e. eGFR < 30 mL/min/ 1.73m2).
6. In the opinion of the Investigator, progression to death is imminent and inevitable within the next 48 - 72 hours, irrespective of the provision of treatment.
7. In the opinion of the Investigator, progression to mechanical ventilation is imminent and inevitable within the next 24 hours, irrespective of the provision of treatment.
8. Possibility of the patient being discharged from hospital within 24 hours.
9. Concurrent participation in other anti-COVID-19 therapeutic or interventional trials. Patients may, at the discretion of the Investigator, concurrently participate in other non-interventional COVID-19 studies.
10. Prior or concurrent use of experimental antiviral therapy for COVID-19 (see Appendix 2.
11. Prior or concurrent use of any interferons other than the investigational product (see Appendix 2)
12. Other known active infections or other clinical conditions (e.g., severe chronic obstructive pulmonary disease) that contraindicate aerosolized inhalation.
13. Patients with current or prior psychiatric illness, seizure disorders, retinal autoimmune disorders, pre-existing severe cardiovascular disease, or patients with prior transplants.
14. Females who are breast-feeding, lactating, pregnant or intending to become pregnant.
15. The subject has any medical condition that in the opinion of the investigator would compromise subject's safety or compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical deterioration | From enrollment to Day 28
  Proportion of patients requiring mechanical ventilation or that die (defined as WHO categories 6, 7, or 8)

SECONDARY OUTCOMES:
Rate of recovery | From enrollment to Day 28
  Proportion of patients demonstrating clinical improvement (defined as WHO categories 0, 1, 2, or 3)
Hospital discharge rate | At Day 28
  Rate of non-hospitalized alive patients
Mortality rate | At Day 28
  Mortality rate
Duration of hospitalization | Up to Day 28
  Number of days hospitalized
Adverse events | From first dose to Day 56
  Adverse event incidence, type and severity

CONTACTS AND LOCATIONS:
Locations (88):
- Argentina (9):
  - Hospital Interzonal General de Agudos Dr Jose Penna, Bahía Blanca
  - Clinica Zabala, Buenos Aires
  - CEMIC, Ciudad Autonoma Buenos Aires
  - Clinica Adventista Belgrano, Ciudad Autonoma Buenos Aires
  - Hospital San Roque, Córdoba
  - Sanatorio del Salvador Privado S.A., Córdoba
  - Sanatorio Privado Duarte Quiroz De Clinica Colombo SA, Córdoba
  - Instituto Medico Rio Cuarto, Río Cuarto
  - Clinica Central S.A., Villa Regina
- Brazil (16):
  - HCPA- Hospital de Clínicas de Porto Alegre, Alegre
  - Fundação PIO XII Hospital de Amor de Barretos, Barretos
  - Hospital Casa de Saúde Vera Cruz (Coordenador), Campinas
  - Hospital São José, Criciúma
  - Hospital das Clínicas UFG, Goiânia
  - Hospital Geral Prof. Dr. Waldemar de Carvalho Pinto Filho de Guarulhos - BR TRIALS, Guarulhos
  - Hospital Felício Rocho, Horizonte
  - Centro de Pesquisas Clínicas da Fundação Doutor Amaral Carvalho, Jaú
  - CePCLIN - Centro de Estudos e Pesquisas em Moléstias Infecciosas, Natal
  - Hospital São Luiz de Jabaquara, Porto Alegre
  - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital 9 de Julho, São Paulo
  - Hospital São Luiz de Jabaquara, São Paulo
  - Instituto de Moléstias Cardiovalsculares Tatuí Ltda, Tatuí
  - Lobus Centro de Pesquisa, Volta Redonda
  - Lóbus Centro de Pesquisa Clínica, Volta Redonda
- Canada (4):
  - University Hospital - London Health Sciences Centre, London
  - Victoria Hospital -London Health Sciences Centre, London
  - St Paul's Hospital, Vancouver
  - St. Boniface Hospital, Winnipeg
- Chile (2):
  - Hospital Base Osorno, Osorno
  - Hospital Sotero del Rio, Santiago
- Colombia (6):
  - Fundacion Cardiovascular de Colombia - Instituto del Carazon Floridablanco, Floridablanca, Santander Department
  - Clinica de la Costa Ltda, Barranquilla
  - Fundacion Hospital Universidad del Norte, Barranquilla
  - Fundacion Oftalmologica, Floridablanca
  - Clinica SOMER, Medellín
  - Corporacion Clinica, Villavicencio
- Indonesia (4):
  - RS Universitas Udayana, Bali
  - Royal Taruma Hospital, Jakarta
  - M. Djamil Hospital, Padang
  - Sardjito Hospital, Yogyakarta
- Kenya (5):
  - KEMRI Kericho, Kericho
  - KEMRI/CGHR Siaya Clinical Research Annexe, Kisumu
  - Victoria Biomedical Research Institute, Kisumu
  - CREATES - Strathmore University Medical Centre, Nairobi
  - Kenyatta National Hospital, Nairobi
- Malaysia (4):
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Miri, Miri
  - Sunway Medical Centre, Petaling Jaya
  - HPUPM, Serdang
- Peru (4):
  - Centro Medico Naval Cirujano Mayor Santiago Tavara, Callao
  - Hospital III Daniel Alcides Carrion - Red Essalud de Tacna, Lima
  - Hospital Nacional Dos de Mayo, Lima
  - Hospital Nacional Arzobispo Loayza, Lima Cercado
- South Africa (10):
  - Tiervlei Trial Centre, Cape Town
  - Tread Research, Cape Town
  - Johese Clinical Research: Unitas, Centurion
  - Drs Sarvan and Moodley, Durban
  - TASK Eden, George
  - MERC SiReN, Johannesburg
  - Nelson Mandela Academic Clinical Research Unit (NeMACRU), Mthatha
  - Into Research, Pretoria
  - Dr JM Engelbrecht Trial Site, Somerset West
  - Clinical Projects Research SA (PTY) LTD, Worcester
- Turkey (Türkiye) (12):
  - Ankara City Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Dicle University, Medical Faculty, Diyarbakır
  - Acibadem Atakent Hospital, Istanbul
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Kartal Lutfi Kirdar Research and Training Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kayseri City Hospital, Kayseri
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Selcuk Universitesi Selcuklu Tip Fakultesi Hastanesi, Konya
  - Ondokuz Mayis Univ. Med. Fac., Samsun
  - Karadeniz Tecnical Uni. Med. Fac., Trabzon
- Ukraine (12):
  - CI Dnipropetrovsk CCH #6 of DRC Dept of Therapy (with pulmonological beds) SI DMA of MoHU, Dnipro
  - CNE CCH #16 of Dnipro City Council, DSMU, Ch of Intern Med #1, Dnipro
  - CNE Ivano-Frankivsk Reg Clin Infectious Hospital of Ivano-Frankivsk Regional Council, Ivano-Frankivsk
  - CNE of Kharkov RC Reg Cl Infectious Hospital, Kharkiv
  - Communal Non-Commercial Medical Enterprise "O.T.Bohayevskyi Kremenchuk City Hospital #1", Kremenchuk
  - Kyiv Municipal Clinical Hospital #17 O. O. Bogomolets NMU, Kyiv
  - City Hospital #1, Mykolaiv
  - City Clinical infectious Hospital, Odesa
  - Poltava Regional Clinical Infectious Hospital Dept of Diagnostics HSEIU Ukrainian Medical Stomatolog, Poltava
  - Municipal Non-Profit Enterprise Central City Hospital Of Rivne City Council, Rivne
  - CCH #1 Vinnytsia M.I.Pyrogov NMU Ch of Infectious Diseases, Vinnytsia
  - CI Central City Hospital #1 of Zhytomyr, Zhytomyr

IPD SHARING:
Plan to Share IPD: Undecided